CLINICAL TRIAL: NCT06367829
Title: Comparing Mortality, Revision Rates, and Patient-Reported Outcomes With Different Stem Lengths of the Lubinus SPII Cemented Hip Stem: A Target Trial Emulation.
Brief Title: Lubinus SPII Hip Stem Target Trial Emulation (LARGE)
Acronym: LARGE
Status: Enrolling by invitation | Type: Observational
Sponsor: JointResearch (Other)
Collaborators: OLVG (Network); Uppsala University (Other); Göteborg University (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: WO.24.025
Record Dates: First submitted 2024-04-04; First posted 2024-04-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-02

CONDITIONS: Treatment Outcome
MeSH Terms: interventions — Microscopy, Electron, Scanning Transmission

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary hip replacement patients: Patients who have received primary hip replacement therapy with an indication of osteoarhritis, osteonecrosis or fracture.
  Interventions: Procedure: Lubinus SPII hip stem 130mm; Procedure: Lubinus SPII hip stem 150mm

INTERVENTIONS:
Procedure: Lubinus SPII hip stem 130mm — Shorter length of the SPII hip stem
  Other Names: 130mm stem
Procedure: Lubinus SPII hip stem 150mm — Longer length of the SPII hip stem
  Other Names: 150mm stem

SUMMARY:
The research questions this study aims to answer are as follows:

Primary research question:

"Do primary total hip arthroplasties for patients with OA, hip fracture or osteonecrosis with the 150mm Lubinus SPII hip stem have better mortality and stem revision rates than primary total hip arthroplasties with the 130mm hip stem?"

Secondary aims include:

* How does line-to-line cementation, compare to undersized cementation in primary total hip arthroplasty for patients with OA, hip fracture, or osteonecrosis when comparing equal size Lubinus SPII hip stems implanted with different cementation techniques?
* Does the Lubinus SPII 150mm hip stem perform equal to the Lubinus SPII 130mm hip stem in primary total hip arthroplasties for patients with OA, hip fracture or osteonecrosis when comparing patient reported outcome measures?

To answer these questions, this study has been allowed use of registered data from the LROI (dutch arthroplasty registry) and the SAR (swedish arthroplasty registry). After exclusion of patients who did not meet inclusion criteria between 2007-2020, approximately 110000 patients remain eligible for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Listed in registry for primary hip arthroplasty.

  * Listed in registry with an indication of osteoarthritis, osteonecrosis or hip fracture.
  * Received the Lubinus SPII hip stem, 130mm or 150mm, for their primary hip arthro- plasty.
  * End point listed in registry (Alive, Deceased or revision).

Exclusion Criteria:

* Patients who received the Lubinus SPII 150 XL conus stem.

Ages: 5 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients incorporated in the LROI and SAR databases between 2007 and 2020 were included, if they satisfied the in- and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 110000 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | From date of surgery to date of event (death), minimally 2 years up to 16 years (2007-2023)
  Time from primary hip surgery to patient death, per hip stem length
Revision rate | From date of surgery to date of event (revision), minimally 2 years up to 16 years (2007-2023)
  Time from primary hip surgery to implant failure, per hip stem length

SECONDARY OUTCOMES:
NRS pain score | before surgery, 3-6 months after surgery, 12 months after surgery
  pain score for rest and activity, rated 0 - 10 (10 is max pain)
Oxford hip score | before surgery, 3-6 months after surgery, 12 months after surgery
  Hip functionality and pain intensity score , 0 - 60, 60 is max pain/least functionality
EQ - 5D | before surgery, 3-6 months after surgery, 12 months after surgery
  Quality of life measurement based on 5 questions with a score of 0 - 100 (how well does patient experience health, 100 is best)
HOOS - PS | before surgery, 3-6 months after surgery, 12 months after surgery
  Hip functionality, disability and pain test, 5 point liker scale ( 0 - 4), higher score is more functional difficulty
Revision rate | From date of surgery to date of event (death), minimally 2 years up to 16 years (2007-2023)
  Time from primary hip surgery to implant failure, per cementation type
Mortality rate | From date of surgery to date of event (revision), minimally 2 years up to 16 years (2007-2023)
  Time from primary hip surgery to patient death, per cementation type

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Poolman, Prof. Dr., Study Chair — OLVG; Ariena Rasker, MSc, Principal Investigator — Joint research OLVG; Tijs de Koningh, Principal Investigator — Joint research OLVG
Locations (1):
- OLVG, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No